CLINICAL TRIAL: NCT03173066
Title: Ferumoxytol as a Contrast Agent for Pulmonary Magnetic Resonance Angiography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrew Michael Siedlecki, Instructor in Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0430172034
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Ferrosoferric Oxide

STUDY DESIGN:
Intervention Model Description: single-arm, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Patients with a clinical concern for pulmonary embolus but not able to receive iodinated contrast will be enrolled. Ferumoxytol will be administered as a contrast agent in coordination with magnetic resonance angiography to identify patency of the cardiopulmonary vasculature.
  Interventions: Drug: Ferumoxytol

INTERVENTIONS:
Drug: Ferumoxytol — ferumoxytol-enhanced magnetic resonance angiography for the diagnosis of pulmonary embolus
  Other Names: Feraheme

SUMMARY:
This proposal is based on findings from our previous work involving ferumoxytol-enhanced cardiac magnetic resonance angiography. The resolution of the pulmonary vasculature based on our previous imaging protocol was exceptional (PMID: 26786296). In the Partners Healthcare System between January 1, 2014 and January 1, 2015 there were 541 patients evaluated in Partners Healthcare-affiliated hospitals with a diagnosis of pulmonary embolism and acute or chronic kidney disease at the same visit between 01/01/2014 and 01/01/2015. Ventilation perfusion scanning was performed in 201 patients during this same time interval. Up to 63% of these patients in one year did not receive the diagnostic test of choice.

DETAILED DESCRIPTION:
Thromboembolic events in patients with chronic kidney disease are out of proportion to age matched controls occurring 2.34 times more frequently than in non-CKD patients (PMID 19561505). At the same time, patients with kidney disease are not offered the gold standard for pulmonary embolus diagnosis, i.e. CT angiography, for concern of acute dialysis to treat contrast-induced nephropathy. Ventilation perfusion scintigraphy (V/Q) is the preferred diagnostic test for patients with advanced CKD (glomerular filtration rate <30mL/min/m2) and suspicion of pulmonary embolus, but can not be utilized if pulmonary parenchyma contains interstitial edema or alveolar occlusion due to pneumonia. If diagnostic tools for pulmonary embolus are not available, patients are subject to the risk of empiric treatment to avoid life-threatening complications of untreated pulmonary embolus. For those patients with CKD that undergo CT angiography, they are placed at risk of initiating dialysis. If this occurs multiple financial costs are associated with dialysis catheter placement and acute hemodialysis. If a patient instead is evaluated with gadolinium-based contrast modalities, there is the risk of nephrogenic systemic fibrosis and the morbidity associated with this iatrogenic disease process.

Ferumoxytol-enhanced MRI could avoid the risk of iodinated contrast and gadolinium contrast and accelerate the diagnosis and treatment of patients with pulmonary embolus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical suspicion for pulmonary embolus
* estimated glomerular filtration rate (eGFR) <30mL/min/1.73m2
* have been clinically disqualified from the use of iodine-based contrast studies, gadolinium-based contrast studies or nuclear-based detection studies

Exclusion Criteria:

* received ferumoxytol in the previous six months
* anaphylactic reaction to other intravenous iron formulations
* calculated estimated glomerular filtration rate is >50mL/min/1.78m2
* patients on dialysis with no residual renal function
* pregnant women and nursing mothers. Standard screening will be used by
* patients >65 years of age with BMI >45, and/or liver disease (Child-Pugh class C)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary embolus | 1 year
  Detection of pulmonary embolus with ferumoxytol-enhanced magnetic resonance angiography

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Siedlecki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data will be offered in publication supplemental material

REFERENCES:
- [Result] Mukundan S, Steigner ML, Hsiao LL, Malek SK, Tullius SG, Chin MS, Siedlecki AM. Ferumoxytol-Enhanced Magnetic Resonance Imaging in Late-Stage CKD. Am J Kidney Dis. 2016 Jun;67(6):984-8. doi: 10.1053/j.ajkd.2015.12.017. Epub 2016 Jan 16. PMID 26786296